CLINICAL TRIAL: NCT06720675
Title: Use of Ex-vivo Hypotermic Perfusion in Patients with Hepatocellular Carcinoma Candidates for Liver Transplant to Reduce the Incidence of Tumor Recurrence
Brief Title: Ex-vivo Hypotermic Perfusion in Patients with Hepatocellular Carcinoma to Reduce the Incidence of Tumor Recurrence
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: HCC-HOPE_2021
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-10

CONDITIONS: Liver Carcinoma; Liver Transplant; Tumor Recurrence; Hepato Cellular Carcinoma (HCC); Hypothermic Oxygenated Machine Perfusion
Keywords: Ex-vivo machine perfusion; Hepato Cellular Carcinoma - HCC; Liver Transplantation - LT; HCC recurrence after LT; Hypothermic Oxygenated Perfusion - HOPE
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SCS - Static Clod Storage: HCC patients transplanted between January 2016 and 2021, who received liver grafts preserved with SCS and a minimum follow-up of 12 months.
  Interventions: Procedure: Static Cold Storage
- HOPE - Hypothermic Oxynated Perfusion: HCC patients transplanted between January 2016 and 2021, who received liver grafts preserved with HOPE and a minimum follow-up of 12 months.
  Interventions: Procedure: Hypothermic Oxygented Perfusion

INTERVENTIONS:
Procedure: Hypothermic Oxygented Perfusion — HOPE start by flushing the organ at low flow values (30 ml/min) with new oxygenated perfusion fluid (cold Belzer MPS solution) during back-table preparation. Hepatic perfusion was performed through the vein leads to a pressure of 3-5 mmHg. Organ were treated with continuous HOPE until transplant and the perfusion was continuously monitored and data downloaded in a USB memory.
  Groups: HOPE - Hypothermic Oxynated Perfusion
Procedure: Static Cold Storage — Liver grafts are stored in sterile organ bags with cold Belzer or Celsior solution and kept in ice at 4°C.
  Groups: SCS - Static Clod Storage

SUMMARY:
This is a retrospective study of single-center cohorts that involves patients with HCC who underwent liver transplantation between January 2016 and 2021, who received livers preserved with Hypothermic Oxygenated Perfusion (HOPE) or Static Cold Storage (SCS) with a minum follow up of 12 months.

DETAILED DESCRIPTION:
The gold standard treatment for Hepatocellular Carcinoma (HCC) is Liver Transplantation (LT) but, despite its success, it maintains cancer recurrence rates of 16%. Ischemia-reperfusion injury (IRI) is considered a major determinant of the higher rate of HCC recurrence associated with transplantation from ECD donors and/or organs with ischemic damage. In this field, the treatment with Machines Perfusion (MP) of the liver has gained increasing attention in the transplant community as a useful tool to relieve IRI, test the hepatic function before transplantation and potentially reconditioning the marginal organs. The current study aims to show that Hypothermic Oxygenated Perfusion (HOPE) can protect recipients not only from IRI and post-transplant complications but also from tumour recurrence, which appears to be inevitably linked to the quality of the organ. This will be done through the comparison between a retrospective group of patients with HCC who have undergone LT with graft preserved by HOPE and a retrospective group of HCC recipients who received grafts preserved without perfusion, but with Static Cold Storage (SCS) technique.

ELIGIBILITY:
Inclusion Criteria:

* Recipients aged 18 years or older with previous diagnosis of HCC, undergone Liver Transplantation at the Transplant Center of the IRCCS AOUBO between January 2016 and 2021
* Patients who have given informed consent to participate in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HCC patients transplanted between January 2016 and 2021 who received liver grafts preserved with HOPE or SCS and minimum 12 months of follow-up will be included in the study. The diagnosis of HCC was confirmed in accordance with the recommendations of international guidelines issued during the period corresponding to the diagnosis. Of these patients, demographic data, clinical parameters, laboratory data and cancer parameters will be collected, including the number of tumors, size, maximum diameter, total tumor diameter, satellite nodules, microvascular invasion, the grade, classification and stage of the tumour. Donor characteristics and post-transplant clinical data of recipients will be collected too.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Risk of HCC tumour recurrence | From liver transplant to twelve months after LT
  For the purposes of descriptive analyses, categorical variables will be expressed as frequency and percentage; continuous variables will be expressed as mean + standard deviation (SD) or with median and inter-quartile range (IQR) depending on their distributive form. Comparisons between the two groups will be made by means of Chi-Quadro tests or Fisher's test (categorical variables), t-tests or Mann-Whitney tests (means of continuous variables, depending on their type of distribution). Multiple logistic regression models will be used to identify factors associated with the appearance of tumour recurrence, in which the graft preservation method is considered as a risk factor and the main characteristics of recipient and donor are included as potential confounders. Survival analysis using Kaplan-Meier curves, log-rank test and Cox regression will be performed to assess the time between transplantation and recurrence and the factors associated with it.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Ravaioli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

REFERENCES:
- [Background] Dajti G, Germinario G, Prosperi E, Siniscalchi A, Vasuri F, Valente S, Odaldi F, Maroni L, Serenari M, Bertuzzo V, Laurenzi A, Del Gaudio M, Cescon M, Ravaioli M. The role of cold ischemia time and hypothermic perfusion in predicting early hepatocellular carcinoma recurrences after liver transplantation. Artif Organs. 2024 Jun;48(6):619-625. doi: 10.1111/aor.14715. Epub 2024 Jan 25. PMID 38270476